CLINICAL TRIAL: NCT01600391
Title: Visual Cue Training to Improve Walking and Turning After Stroke: a Pilot Study
Brief Title: Visual Cues for Gait Training Post-stroke
Acronym: VCTpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Collaborators: University of Birmingham (Other); University of Nottingham (Other); Stroke Research Network (Unknown); University of Newcastle, Australia (Other)
Responsible Party: Principal Investigator, Dr Kristen Hollands, Chief Investigator, University of Salford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VCTpilot
Record Dates: First submitted 2012-05-10; First posted 2012-05-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Stroke
Keywords: Stroke; Visual cues; Gait rehabilitation; Walking adaptability; Turning; Overground walking; Treadmill training
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Care (Active Comparator): A task specific-based intervention that does not include use of visual cues to influence quality or adaptability of gait.
  Interventions: Behavioral: Usual care
- Overground visual cue training (Experimental): Overground visual cue training will involve stepping to targets which are positioned to improve gait symmetry and speed. Training will include turning practice and the avoidance of obstacles for adaptability during straight walking.
  Interventions: Behavioral: Overground visual cue training
- Treadmill visual cue training (Experimental): Treadmill training with visual cues will be delivered using a force-instrumented treadmill (CMill, Forcelink, NL). Walking training will involve stepping to targets which are positioned to improve gait symmetry and speed. Training will include turning practice and the avoidance of obstacles for adaptability during straight walking.
  Interventions: Behavioral: Treadmill visual cue training

INTERVENTIONS:
Behavioral: Usual care — Walking rehabilitation for 1 hour, 2 times per week and 8 weeks duration. Usual care intervention that does not include use of visual cues to influence quality or adaptability of gait.
  Other Names: Standard care; Standard physiotherapy
  Arms: Usual Care
Behavioral: Overground visual cue training — Walking rehabilitation for 1 hour, 2 times per week and 8 weeks duration. Overground visual cue training will involve stepping to targets, which are positioned to improve walking pattern according to needs identified in baseline assessment. Treatment will progress from practice of improved stepping pattern (symmetry of stepping) and speed to practice of adjusting footfalls by avoiding targets randomly, as one might need to be able to do to avoid an obstacle or an uneven surface. Training will also involve turning practice.Overground visual cue training will be delivered by National Health Service therapists in participating National Health Service sites.
  Other Names: Visual cue gait training
  Arms: Overground visual cue training
Behavioral: Treadmill visual cue training — Walking rehabilitation for 1 hour, 2 times per week and 8 weeks duration. Treadmill training with visual cues will be delivered using a force-instrumented treadmill (CMill, Forcelink, NL). The Treadmill visual cue training will involve participants stepping to targets shone onto a treadmill. Treatment will progress from practice of improved stepping pattern (symmetry of stepping) and speed to practice of adjusting footfalls by avoiding targets randomly, as one might need to be able to do to avoid an obstacle or an uneven surface. Training will also involve turning practice. Treadmill visual cue training will be delivered by qualified physiotherapists at the University of Birmingham.
  Other Names: CMill, Forcelink, NL
  Arms: Treadmill visual cue training

SUMMARY:
Given that visual information comprises one of the most important and salient sources of information used during walking, that visual cues have been shown to be more effective than auditory cues in triggering gait adjustments and that stroke survivors have been reported to become more dependent on visual cues, the investigators hypothesize that visual cues would be more effective in triggering gait recovery and adaptability following stroke than interventions not including visual cues.

The investigators will integrate visual cues with walking and turning practice, and contrast this intervention to routine overground walking practice. Stroke participants recruited from NHS stroke rehabilitation clinics in the West Midlands, will be randomized to one of three gait rehabilitation groups. Each group will receive the same frequency and duration of treatment delivered by qualified physiotherapists. Overground visual cue training (OVCT) and usual care (UC) groups will be treated in participating NHS sites. Treadmill training with visual cues (TVCT) will take place at the University of Birmingham.

DETAILED DESCRIPTION:
The gait of many stroke patients remains impoverished and characterized by impairments including asymmetries in propulsive forces between the paretic and non-paretic limbs, step lengths, widths and stance and swing phase durations. Currently there is insufficient evidence that current rehabilitation strategies improve walking in people who are more than 6 months post-stroke.

The purpose of the trial is to determine the necessary information on which to base a future definitive trial examining the effectiveness of visual cues for gait training following stroke in contrast to conventional over-ground walking practice.

The study will determine the numbers of patients willing to be recruited into both control and VCT groups; the willingness of physiotherapists at each collaborating site to enroll patients to usual care OVCT and TVCT groups.

It will determine the numbers of patients who do not complete the allocated treatment, thus dropping out of the study, and the reasons for dropping out.

The knowledge gathered about recruitment, outcomes and drop-out rates will determine sample size for a subsequent definitive trial.

The study will also measure completeness of outcome data, i.e. percentage of patients with no missing values in outcome assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Able to walk 10 metres with or without assistance
* Residual paresis in the lower limb (Fugl-Meyer Lower Limb score less than 34)
* Informed written consent.

Exclusion Criteria:

* Gait speed more than 0.8 m/s
* Patients with a premorbid (retrospective) modified Rankin Scale score of greater than 3
* Gait deficits attributable to non-stroke pathology
* Visual impairments preventing use of visual cue training (as assessed by Apple Cancellation test
* Concurrent progressive neurologic disorder, acute coronary syndrome, severe heart failure, confirmed or suspected lower-limb fracture preventing mobilization, and those requiring palliative care
* Inability to follow a three step command (as assessed by Modified mini-mental status exam).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Participant enrollment, recruitment and retention. | Ongoing for18 months after start of recruitment.
  Determine:
  1. The numbers of patients willing to be recruited into both control and VCT groups.
  2. The willingness of physiotherapists at each collaborating site to enrol patients to both control and VCT groups.
  3. The numbers of patients who do not complete the allocated treatment, thus dropping out of the study, and determine the reasons for dropping out.
  4. Measure completeness of outcome data, i.e. percentage of patients with no missing values in outcome assessments.

SECONDARY OUTCOMES:
180 degree turn | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  Time taken (s) and number of steps (#) to complete a 180 degree turn
Gait adaptability | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  The number of times participants fail to hit stepping targets when these are presented unpredictably in timing and location will be used to indicate the ability to adapt the straight gait pattern according to environmental demands.
Timed up and Go (TUG) test (7m) | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  The subject begins by sitting up strait in a chair with their hands on their thighs and their backs touching the back of the chair. After they are given the go signal, they rise from the chair, walk at their normal speed, turn around right after passing the tape at the end of the pathway, return back to the chair, turn around and sit down.
Fugl-Meyer Lower Limb Motor Assessment | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  Items are rated on a three point scale (0= cannot perform, 1 = performs partially, 2 = performs fully) and standardised protocols for administration will be followed
Berg Balance Scale | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
Falls Efficacy Scale | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  This will assess changes in confidence to walk without falling which may be expected as a result of practice of adaptable walking
SF-12 | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  This is a short-form health survey with only 12 questions. It yields an 8-scale profile of functional health and well-being scores, including physical functioning, and social, emotional, mental and general health and has been included to measure effects on broader quality of life
Functional ambulation category | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
Gait speed | Assessments take place at baseline, after completion of an 8 week training program and follow up at 3 months
  Proportion of participants achieving a gait speed of 0.4 m/s and 0.8 m/s. Gait speed will be measured during a 10 metre walk.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hollands, PhD, Principal Investigator — University of Salford
Locations (4):
- United Kingdom (4):
  - Birmingham Community Health Care NHS Trust, Birmingham, West Midlands
  - Sandwell and West Birmingham Hopsitals NHS Trust, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - South Warickshire NHS Foundation Trust, Birmingham

REFERENCES:
- [Background] Aziz NA, Leonardi-Bee J, Phillips M, Gladman JR, Legg L, Walker MF. Therapy-based rehabilitation services for patients living at home more than one year after stroke. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD005952. doi: 10.1002/14651858.CD005952.pub2. PMID 18425928
- [Background] Bank PJ, Roerdink M, Peper CE. Comparing the efficacy of metronome beeps and stepping stones to adjust gait: steps to follow! Exp Brain Res. 2011 Mar;209(2):159-69. doi: 10.1007/s00221-010-2531-9. Epub 2011 Jan 8. PMID 21221956
- [Background] Bonan IV, Yelnik AP, Colle FM, Michaud C, Normand E, Panigot B, Roth P, Guichard JP, Vicaut E. Reliance on visual information after stroke. Part II: Effectiveness of a balance rehabilitation program with visual cue deprivation after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2004 Feb;85(2):274-8. doi: 10.1016/j.apmr.2003.06.016. PMID 14966713
- [Background] Patla AE. Understanding the roles of vision in the control of human locomotion. Gait and Posture 5,(1):54-69,February 1997.
- [Background] Lehmann JF, Condon SM, Price R, deLateur BJ. Gait abnormalities in hemiplegia: their correction by ankle-foot orthoses. Arch Phys Med Rehabil. 1987 Nov;68(11):763-71. PMID 3675173
- [Background] Griffin MP, Olney SJ et al. Role of symmetry in gait performance of stroke subjects with hemiplegia. Gait and Posture 3: 132-142, 1995
- [Background] Barela JA, Whitall J, et al. An examination of constraints affecting the intralimb coordination of hemiparetic gait. Human Movement Science 19: 251-273, 2000.
- [Background] Hollands MA, Patla AE, Vickers JN. "Look where you're going!": gaze behaviour associated with maintaining and changing the direction of locomotion. Exp Brain Res. 2002 Mar;143(2):221-30. doi: 10.1007/s00221-001-0983-7. Epub 2002 Jan 10. PMID 11880898
- [Derived] Hollands KL, Pelton TA, Wimperis A, Whitham D, Tan W, Jowett S, Sackley CM, Wing AM, Tyson SF, Mathias J, Hensman M, van Vliet PM. Feasibility and Preliminary Efficacy of Visual Cue Training to Improve Adaptability of Walking after Stroke: Multi-Centre, Single-Blind Randomised Control Pilot Trial. PLoS One. 2015 Oct 7;10(10):e0139261. doi: 10.1371/journal.pone.0139261. eCollection 2015. PMID 26445137
- [Derived] Hollands KL, Pelton T, Wimperis A, Whitham D, Jowett S, Sackley C, Alan W, van Vliet P. Visual cue training to improve walking and turning after stroke: a study protocol for a multi-centre, single blind randomised pilot trial. Trials. 2013 Sep 3;14:276. doi: 10.1186/1745-6215-14-276. PMID 24004882